CLINICAL TRIAL: NCT04216693
Title: Efficacy and Safety of Digoxin in the Treatment of Adults Patients With Non-alcoholic Steatohepatitis: a Multi-center, Randomized, Placebo-controlled Trial
Brief Title: Digoxin for Patients With Non-alcoholic Steatohepatitis (NASH)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative decision to terminate.
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Beicheng Sun, Professor; Director of the department of hepatobiliary surgery; Doctor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: v1.0 20200101
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-07

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic Steatohepatitis; Digoxin; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digoxin tablet (Experimental): Patients will be given digoxin orally daily for 24 weeks. The initial dose will be selected with the goal of achieving a serum digoxin concentration of 0.7-1 ng/ml, a dose range recommended for heart failure patients. A dose of 0.0625, 0.125 or 0.25 mg daily will be selected based on a normogram.
  Interventions: Drug: Digoxin tablet
- Placebo (Placebo Comparator): Digoxin-like oral placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Digoxin tablet — The NASH patients in experimental group will take digoxin tablets orally with the goal of achieving a serum digoxin concentration of 0.7-1 ng/ml for 24 weeks.
  Arms: Digoxin tablet
Other: Placebo — The control group will receive the digoxin-like placebo treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess if digoxin is safe and efficacious in treating patients with non-alcoholic steatohepatitis (NASH) within the approved target range of 0.7 to 1 ng/ml.

DETAILED DESCRIPTION:
This study is a phase II, open labeled, multi-center, prospective, randomized, placebo controlled clinical trial to evaluate the efficacy and safety of digoxin in the treatment of nonalcoholic steatohepatitis. The participants will take study drug digoxin, which is approved by FDA for the treatment of congestive heart failure (CHF), orally daily based on the body weight, titrated to the level of 0.7 to 1 ng/ml for total of 6 cycles (4 weeks/cycle). A liver biopsy will be performed at the beginning of the study and 24 weeks after randomization to evaluate the efficacy of digoxin in the treatment of nonalcoholic steatohepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to voluntarily sign an informed consent form (ICF) and Health Insurance Portability and Accountability Act (HIPAA) authorization.
2. Males or females between 18-70 years old with a clinically confirmed diagnosis of NASH within the last 12 months of Screening Visit.
3. BMI between 25 and 45 kg/m2.
4. Negative urine drugs-of-abuse screen.
5. Negative alcohol screen.
6. Negative urine pregnancy test and agree to use a medically acceptable method of contraception throughout the study and for 1 month after completing the study. Medically acceptable methods of contraception that may be used by the subject and/or partner include, but are not limited to: abstinence, oral contraception, NuvaRing® or transdermal systems, diaphragm with vaginal spermicide, intra uterine device, condom and partner using vaginal spermicide, at least 6 months after surgical sterilization, progestin implant or injection, or postmenopausal female (no menstrual period for > 2 years) or vasectomy (>6 months).
7. Normal EKG.
8. Deemed normal age-adjusted creatinine level.
9. NAS score greater than 5.
10. Steatosis greater than 8% on liver biopsy. Able and willing to comply with the protocol and available for all scheduled clinic visits and telephone calls.

Exclusion Criteria:

1. Known cardiovascular disease
2. Subjects who have previously received digoxin or who have history of hypersensitivity, allergy, intolerance or contraindication to digoxin.
3. Requiring any of the following medications during the duration of the study:

   * Potassium-depleting diuretics
   * Calcium, particularly if administered rapidly by the intravenous route
   * Quinidine, verapamil, amiodarone, propafenone, indomethacin, itraconazole, alprazolam, erythromycin, clarithromycin (and possibly other macrolide antibiotics), tetracycline, propantheline, diphenoxylate, antacids, kaolin-pectin, sulfasalazine, neomycin, cholestyramine, certain anticancer drugs, metoclopramide, rifampin, quinine, penicillamine, thyroid hormone, sympathomimetics. Succinylcholine, calcium channel blockers, beta-blockers, carvedilol, and any drug that may cause a significant deterioration in renal function.
4. History of cirrhosis based on imaging or clinical criteria and/or hepatic decompensation including ascites, hepatic encephalopathy or variceal bleeding.
5. Platelet count < 100,000/ul
6. Albumin below 3.5 g/dl
7. Serum ferritin > 800 ng/mL
8. Anti-neutrophil antibody above 1: 160
9. International normalized ratio (INR) > 1.2History of liver transplantation
10. History of hepatocellular carcinoma (HCC)
11. History of malignancy within the past 5 years or ongoing malignancy other than basal cell carcinoma, or resected noninvasive cutaneous squamous carcinoma at the time of Screening visit
12. Active, serious infections that requires parenteral antibiotic or antifungal therapy within 30 days prior to Screening visit.
13. Any ≥Grade 3 laboratory abnormality as defined by Toxicity Grading Scale, with the following exceptions unless clinical assessment foresees an immediate health risk to the subject:

    * Subjects with pre-existing diabetes or with asymptomatic glucose ≥Grade 3 elevations;
    * Subjects with asymptomatic triglyceride or cholesterol ≥Grade 3 elevations;
    * Subjects with asymptomatic ALT and/or AST > 4 time above normal
14. Females who are pregnant or breastfeeding.
15. Current or anticipated treatment with radiation therapy, cytotoxic chemotherapeutic agents and immunomodulating agents (such as systemic corticosteroids, interleukins, interferons).
16. Use of any experimental medications within the last 6 months of Screening Visit.
17. Any other clinically significant disorders or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing and protocol requirements.
18. Familial dyslipidemia.
19. Weight loss of >5% within 6 months prior to Screening, based on subject's reporting
20. Currently or participated in a weight loss program within the last 6 months.
21. Any history of bariatric surgery.
22. Diabetes mellitus Type I
23. Daily alcohol intake >20 ml (2 units)/day for women and 30 ml (3 units)/day for men (on average), as per Alcohol Use Disorders Identification Test (AUDIT) questionnaire at Screening and plan to consume the same alcohol amount referenced above during the trial.
24. Hemoglobin A1c >9.0%
25. Treatment initiation or dose change within 3 months of Screening with Vitamin E, or any of the following anti- diabetic medications: DPP-4 inhibitor, GLP-1 receptor agonists (such as Januvia [sitagliptin], Byetta [incretin], etc.), pioglitazone, or SGLT2 inhibitors ("gliflozin" drugs), Metformin, fibrates, statins, insulin, Vitamin D, or sulfonylurea.
26. Use of any immunosuppressive medication, anti-inflammatory monoclonal antibody treatment, or chronic systemic corticosteroids >10 mg prednisone-equivalent concurrently or within 1 year prior to Screening.
27. Uncontrolled or clinically unstable thyroid disease, in the judgment of the Principal Investigator.
28. History or presence of hepatitis B or C or human immunodeficiency virus (HIV).
29. Uncontrolled arterial hypertension
30. Any severe, acute, or chronic medical or psychiatric condition that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Two point change in histological NAFLD activity score (NAS) | Baseline, 24 weeks
  Non-alcoholic fatty liver disease score (NAS) is a histological classification to assess the severity of liver steatosis, lobular inflammation and ballooning in the liver biopsy, which ranges from 0-8 with the increase in number representing a worse outcome. Therefore, the efficacy improvement was to be at least 2 points in lowering the score.
Proportion of subjects with at least a 30% change in % steatosis relative to screening | Baseline, 24 weeks
  Liver steatosis is graded based on the percentage of fat within the hepatocytes: grade 0 (healthy, <5%), grade 1 (mild, 5%-33%), grade 2 (moderate, 34%-66%), and grade 3 (severe, >66%). the efficacy improvement was to be proportion of subjects with at least a 30% decrease in % steatosis relative to screening.

SECONDARY OUTCOMES:
Change in the mean concentration of serum aspartate aminotransferase (AST) | 0, 2, 4, 6, 11, 24 weeks
Change in the mean concentration of serum alanine aminotransferase (ALT) | 0, 2, 4, 6, 11, 24 weeks
Change in liver histological fibrosis staging | Baseline, 24 weeks
  Fibrosis staging was measured as following criteria: 0=none, 1=perisinusoidal or periportal fibrosis, 2=perisinusoidal and portal/periportal fibrosis, 3=bridging fibrosis, and 4=cirrhosis.the definition of fibrosis stages improvement requires at least one stage.

OTHER OUTCOMES:
Change in the mean concentration of serum inflammation markers | 0, 2, 4, 6, 11, 24 weeks
  Change from baseline in Interleukin (IL)-6, C-reactive Protein (CRP).

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ouyang X, Han SN, Zhang JY, Dioletis E, Nemeth BT, Pacher P, Feng D, Bataller R, Cabezas J, Starkel P, Caballeria J, Pongratz RL, Cai SY, Schnabl B, Hoque R, Chen Y, Yang WH, Garcia-Martinez I, Wang FS, Gao B, Torok NJ, Kibbey RG, Mehal WZ. Digoxin Suppresses Pyruvate Kinase M2-Promoted HIF-1alpha Transactivation in Steatohepatitis. Cell Metab. 2018 Feb 6;27(2):339-350.e3. doi: 10.1016/j.cmet.2018.01.007. PMID 29414684